CLINICAL TRIAL: NCT05678400
Title: Comparison of the Immediate Effects of a Hypopressive Abdominal Exercise Program Versus a Proprioceptive Neuromuscular Facilitation Stretching Program on Hamstring Flexibility in Adults With Short Hamstring Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Associate professor in health sciences, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Andres TFM
Record Dates: First submitted 2023-01-02; First posted 2023-01-10 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Exercise Therapy; Physical Therapy Modalities; Hamstring Muscles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypopressive abdominal techniques (Experimental): All subjects were instructed by a registered physiotherapist on how to correctly perform the hypopressive abdominal techniques (HAT) in two familiarisation sessions of 45 minutes each before any action was taken. After the two sessions, all subjects who did not learn the exercise correctly were dropped from the study. The HAT training consisted of asking subjects in a standing position to perform a spinal elongation with neutral pelvis and scapular muscle activation for three normal respiratory cycles with slow and deep exhalation, and on the last breath, an expiratory apnoea with rib expansion and elevation was requested. In this session, following the guidelines described in the familiarisation sessions, two series of four dynamic HATs in standing position were performed: dynamic HATs in right tilt, dynamic HATs in left tilt, dynamic HATs in right rotation and dynamic HATs in left rotation.
  Interventions: Behavioral: Hypopressive abdominal techniques
- Stretching of proprioceptive neuromuscular facilitation (Active Comparator): The therapist straddled that leg, and raised the other leg by placing the heel on the shoulder. The therapist then flexed the participant's hip, maintaining knee extension, to the point of discomfort indicated by the patient or the therapist's perceived end of range. In this position the leg was held straight for 10 seconds and immediately afterwards the participant was asked to perform a maximum isometric contraction for 5 seconds using the therapist's shoulder as counter resistance, thus keeping the leg straight at the same point. As soon as the contraction stops, the therapist flexes the hip again until a new range limit is reached, repeating the same protocol again. The total duration is 60 seconds, consisting of 4 passive stretches of 10 seconds each and 4 isometric contractions against resistance of 5 seconds each.
  Interventions: Behavioral: Stretching of proprioceptive neuromuscular facilitation

INTERVENTIONS:
Behavioral: Hypopressive abdominal techniques — Both training protocols were carried out in a single intervention for each of the participants assigned to either the HAT or the PNF stretching group. The intervention began with the measurement of hip flexion using the EPR test, and ended with a post-intervention measurement of hip flexion to observe the effects of the treatment. All measurements, as well as the interventions for each of the patients in the two groups, were carried out by the same registered physiotherapist. In order to standardise an order of examination of the lower limbs in the EPR test, the right lower limb was assessed first, followed by the left lower limb. Likewise, the same order was standardised for stretching in the PNF group.
  Arms: Hypopressive abdominal techniques
Behavioral: Stretching of proprioceptive neuromuscular facilitation — Stretching of proprioceptive neuromuscular facilitation
  Arms: Stretching of proprioceptive neuromuscular facilitation

SUMMARY:
A Randomised Controlled Trial was conducted to assess increases in hamstring flexibility using two different methods, one group of participants who were stretched with PNF techniques and the other group who performed Hypopressive Abdominal Techniques (HAT). Flexibility scores of both groups were obtained and compared using pre and post measurements of a single intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants with less than 75° in the straight leg raise test.

Exclusion Criteria:

* History of hamstring injury within the last year.
* Pharmacological treatment or history of neurological, orthopaedic, growth or autoimmune disorders.
* Training to improve flexibility in the week prior to the intervention.
* Hypertension.
* Pregnant women.
* Inability to perform hypopressive abdominal techniques.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-26 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Straight leg raise test. | Baseline changes at the end of the intervention (approximately one hour).
  The subject in supine decubitus. The patient's unscanned leg was kept stretched out on the stretcher by means of thigh straps. A digital inclinometer was placed on the other leg over the tibia before starting to lift the leg, in order to be able to quantify the degrees obtained during the test. The therapist will place one hand on the patient's heel holding the calcaneus to prevent rotation and the other on the patella to prevent the knee from flexing during the test. The examiner shall then perform a slow, progressive flexion of the hip with the knee extended, starting from 0° at rest and considering 90° when the lower limb is completely perpendicular to the examination couch. The angular value is taken as the maximum degree of flexion tolerated by the individual, the moment at which the pelvis begins to tilt in retroversion or when the examiner perceives a feeling of firm resistance.

SECONDARY OUTCOMES:
The Toe-Floor Distance test | Baseline changes at the end of the intervention (approximately one hour).
  The Toe-Floor Distance test was also used as a tool to measure the flexibility of the hamstring muscles. The subject stood on a platform without shoes and with feet hip-width apart. The subject was asked to lean forward, flexing the trunk as far as possible, keeping the knees, arms and fingers fully extended. The vertical distance between the tip of the middle finger and the platform was measured with a flexible tape measure and expressed in centimetres. The vertical distance between the platform and the tip of the middle finger was positive when the subject did not reach the platform and negative when the subject could reach further.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultade de fisioterapia, Pontevedra, Spain